CLINICAL TRIAL: NCT04947241
Title: Phase Ib Clinical Study of Toripalimab Combined With Gemcitabine and Cisplatin Neoadjuvant Chemotherapy in Patients With Resectable Locally Advanced Head and Neck Squamous Cell Carcinoma
Brief Title: Toripalimab Combined With Gemcitabine and Cisplatin Treating Resectable Locally Advanced HNSCC
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Zhigang Liu, Chief physicion, Fifth Affiliated Hospital, Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: No.ZDWY[2020]LunziNo.(K66-1)
Record Dates: First submitted 2021-06-18; First posted 2021-07-01 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Locally Advanced Head and Neck Squamous Cell Carcinoma; Neoadjuvant Therapy
Keywords: Anti-PD-1 Monopoly Antibody; immunochemotherapy; head and neck squamous cell carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Cisplatin; toripalimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant therapy (Experimental): Patients included are going to receive neoadjuvant therapy, surgery and adjuvamt therapy post surgery. Before surgery, patients will receive therapy as follows: PD-1 inhibitor: 240mg (day1) , intravenous, Q3W, 2cycles; cisplatin: 80 mg/m2(day1), intravenous , intravenous, Q3W, 2cycles Gemcitabine: 1000mg/m2(day1and day8), intravenous, Q3W, 2cycles
  Interventions: Drug: PD-1 inhibitor+ Gemcitabine + Cisplatin

INTERVENTIONS:
Drug: PD-1 inhibitor+ Gemcitabine + Cisplatin — Before surgery, patients will receive therapy as follows:
  PD-1 inhibitor: 240mg (day1) , intravenous, Q3W, 2cycles; cisplatin: 80 mg/m2(day1), intravenous , intravenous, Q3W, 2cycles Gemcitabine: 1000mg/m2(day1and day8), intravenous, Q3W, 2cycles
  Other Names: Toripalimab

SUMMARY:
Head and Neck Squamous Cell Carcinoma (HNSCC) is the most common malignant tumor of the head and neck, accounting for 90% of head and neck malignancies, and 16% to 40% of systemic malignancies. There are 60,000 new cases reported annually worldwide, and the incidence and mortality are increasing year by year, however,the 5-year survival rate under standard treatment is only 50%. 70%~80% of patients already developed into locally advanced status (stage II-IVa) when they are first diagnosed. The treatment principle is mainly determined by the clinical stage and location of the tumor, various factors affecting the prognosis and the patient's tolerance. Locally advanced head and neck squamous cell carcinoma has a higher probability of local/regional failure and distant metastasis after treatment. Therefore, in recent years, the use of neoadjuvant therapy (NAC) followed by surgery or radiotherapy has been advocated. Surgical treatment is still one of the preferred treatments for local head and neck squamous cell carcinoma. TPF (Docetaxel + Cisplatin + Fluorouracil) regimen is considered as the standard regimen of induced chemotherapy for head and neck squamous cell carcinoma (especially in laryngeal cancer), which can significantly reduce the patient's distant metastasis rate and prolong overall survival ( OS). Nevertheless, the therapeutic effect of neoadjuvant therapy on head and neck squamous cell carcinoma has reached a bottleneck. In recent years, PD-1 inhibitors have achieved significant effects in the field of tumor therapy and have been approved for the treatment of various tumors including head and neck tumors. And a number of clinical trials have shown that PD-1 inhibitors can significantly prolong the OS of patients.

Altogether, the investigators launch an open-label, single-arm, phase Ib clinical trial of PD-1 inhibitor plus chemotherapy in patients with resectable HNSCC to explore the safety and efficacy of the treatment. The study comprises two stages, run-in and case development.

DETAILED DESCRIPTION:
In the first phase, we would observe the initial six patients lasting 90 days from the first day of treatment(or 30 days after surgery) to evaluate if the dose-limited- toxicity DLT would occur in two of them or more.

3、If the dose-limited- toxicity would be recorded in no more than one patient, the trail would continue until meeting the scheduled size of population, otherwise the trial would stop. The further investigation would be launch to review the data thoroughly and modify the protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Untreated locally advanced head and neck squamous cell carcinoma confirmed by histology or cytology;
2. Patients who are recommended to perform surgery;
3. Patients between 18 and 70 years old;
4. ECOG: 0～2 points;
5. Estimated survival time ≥ 6 months;
6. At least one measurable lesion should be detected according to the RECIST 1.1;
7. The major organs meet the following standards (no blood components and cell growth factors are injected within 14 days):

   1. Hemoglobin HB≥90 g/L; neutrophil ANC≥1.5×109/L; platelet count PLT≥100×109/L;
   2. Serum albumin ≥28g/L;
   3. Total bilirubin TBIL≤1.5×upper limit of normal, alanine aminotransferase ALT, aspartate aminotransferase AST≤2.5×upper limit of normal; if there is liver metastasis, ALT and AST≤5×upper limit of normal;
   4. Serum creatinine ≤1.5×upper limit of normal, and creatinine clearance ≥50 mL/min;
   5. Activated partial thromboplastin time (APTT) and international normalized ratio (INR) ≤ 1.5 × upper limit of normal (for the use of stable doses of anticoagulant therapy such as low molecular weight heparin or warfarin, and INR in the anticoagulant expected treatment can be filtered within the scope);
   6. TSH≤ upper limit of normal; if abnormal, the T3 and T4 levels should be examined, and the T3 and T4 levels are normal.
8. Women of childbearing age should take contraceptive measures (such as intrauterine devices, contraceptives or condoms) during the medication period and within 3 months after the medication; the serum or urine pregnancy test is negative within 7 days before the study is enrolled, And must be a non-lactating patient, and the male should agree to take contraceptive measures during the study period and within 3 months after the end of the study period;
9. The subjects voluntarily joined the study, signed an informed consent form, had good compliance, and cooperated with the follow-up.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Allergic to anti-PD-1 monoclonal antibody, gemcitabine, or cisplatin;
3. History of other malignant tumors in the past 5 years or at the same time, except for cured skin basal cell carcinoma, cervical carcinoma in situ, and thyroid papillary carcinoma;
4. Uncontrollable clinical symptoms or diseases of the heart, such as: (1) Heart failure, NYHA Ⅱ, III or IV (2) Unstable angina (3) Myocardial infarction occurred within 1 year (4) Supraventricular in clinical significance or Patients with ventricular arrhythmia requiring clinical intervention;
5. Have received any of the following treatments:

   1. Have received any research relevant drugs before enrolling in this research;
   2. Enrolled in another clinical study at the same time, unless it is an observational (non-interventional) clinical study or intervention in a new clinical study follow-up;
   3. Patients who need to be given corticosteroids (more than 10 mg prednisone equivalent dose per day) or other immunosuppressive agents for systemic treatment within 2 weeks before giving medication for the first time, except for local inflammation and prevention of allergies, nausea and vomiting The case of corticosteroids. In the absence of active autoimmune diseases, inhaled or topical steroids and adrenal corticosteroids with a dose greater than 10 mg per day of prednisone curative dose are allowed to replace;
   4. Have been vaccinated with anti-tumor vaccine or have been vaccinated with live vaccine within 4 weeks before the first administration of study drug;
   5. Received major surgery or severe trauma within 4 weeks before using the study drug for the first time;
   6. The left ventricular ejection fraction of the heart is greater than or equal to 60%;
6. Severe infection (CTC AE greater than grade 2) occurred within 4 weeks before the first use of the study drug, such as severe pneumonia, bacteremia, infection comorbidities that require hospitalization, etc.; baseline chest imaging examinations suggest active lung inflammation , There are symptoms and signs of infection 2 weeks before the first use of the study drug or the need for oral or intravenous antibiotic treatment (excluding prophylactic use of antibiotics);
7. Have active autoimmune diseases, history of autoimmune diseases;
8. A history of immunodeficiency, including a positive HIV test, or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation and bone marrow transplantation;
9. Patients with active tuberculosis infection found through medical history or CT examination, or patients with a history of active tuberculosis infection within 1 year before enrollment, or patients with a history of active tuberculosis infection but without formal treatment 1 year before being checked;
10. The subject has active hepatitis (HBV DNA ≥ 2000IU/ml or 10,000 copies/ml), hepatitis C (hepatitis C antibody is positive, and HCV-RNA is higher than the lower limit of the analysis method);
11. History of psychotropic drug abuse, alcohol and drug abuse;
12. Symptomatic brain metastases (confirmed or suspected);
13. The patients who are reckoned as not suitable for inclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Major pathological response rate | 1 week after surgery
  The proportion of patients with less than 10% surviving cancer cells
Objective Response Rate | 1 week after surgery
  The proportion of patients whose tumors have shrunk to a certain amount and maintained for a certain period of time, including complete response and partial response
R0 resection rate | 1 week after surgery
  The proportion of no residue on the edge of the resection under the microscope after surgery
the incidence of adverse event | 90 days from the first day of treatment
  the immune limited adverse event

SECONDARY OUTCOMES:
Progression Free Survival | 1 year after therapy
  The period of time between the start of treatment for patients with tumor disease and the observation of disease progression or death from any cause
Progression Free Survival | 3 years after therapy
  The period of time between the start of treatment for patients with tumor disease and the observation of disease progression or death from any cause
Progression Free Survival | 5 years after therapy
  The period of time between the start of treatment for patients with tumor disease and the observation of disease progression or death from any cause
Overall Survival | 1 year after therapy
  The time from the start of treatment to death for any cause
Overall Survival | 3 years after therapy
  The time from the start of treatment to death for any cause
Overall Survival | 5 years after therapy
  The time from the start of treatment to death for any cause
Disease Free Survival | 1 year after therapy
  The time from the start of treatment to the first tumor recurrence/metastasis or the death of the patient for any reason
Disease Free Survival | 3 years after therapy
  The time from the start of treatment to the first tumor recurrence/metastasis or the death of the patient for any reason
Disease Free Survival | 5 years after therapy
  The time from the start of treatment to the first tumor recurrence/metastasis or the death of the patient for any reason

CONTACTS AND LOCATIONS:
Overall Officials: Zhigang Liu, M.D., Principal Investigator — Fifth Affilliated Hospital of Sun Yat-sen University
Locations (1):
- Fifth Affilliated Hospital of Sun Yat-sen University, Zhuhai, Guangdong, China